CLINICAL TRIAL: NCT03215498
Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of Faster-acting Insulin Aspart When Administered as a Bolus in a Continuous Subcutaneous Infusion Regimen in Subjects With Type 1 Diabetes
Brief Title: A Research Study of How Faster-acting Insulin Aspart Moves Into, Through, and Out of the Body and How it Works in the Body When Given Through an Insulin Pump to People With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1218-4349; 2016-004306-34 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1189-1545 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-06-29; First posted 2017-07-12 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Faster aspart followed by insulin aspart (Experimental): Each participant will have 2 dosing visits (faster aspart and insulin aspart), the order decided by lottery
  Interventions: Drug: Faster-acting insulin aspart; Drug: Insulin aspart
- Insulin aspart followed by faster aspart (Experimental): Each participant will have 2 dosing visits (faster aspart and insulin aspart), the order decided by lottery
  Interventions: Drug: Faster-acting insulin aspart; Drug: Insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — In a euglycaemic clamp setting each participant will receive a priming dose of 0.08 U/kg body weight, followed by a continuous basal rate of 0.02 U/kg body weight/h and finally a bolus dose of 0.15 U/kg body weight on top of the basal rate
Drug: Insulin aspart — In a euglycaemic clamp setting each participant will receive a priming dose of 0.08 U/kg body weight, followed by a continuous basal rate of 0.02 U/kg body weight/h and finally a bolus dose of 0.15 U/kg body weight on top of the basal rate

SUMMARY:
The aim of the study is to compare the pharmacokinetics (i.e. the course of the blood concentrations of the administered trial drug) of faster-acting insulin aspart (faster aspart), and the currently marketed formulation of insulin aspart (NovoRapid®) when given as a bolus using an insulin pump in people with type 1 diabetes. The pharmacodynamic response (i.e. the course of the blood sugar lowering effect of the administered trial drug) and the safety and tolerability of faster aspart and NovoRapid® will also be assessed.

The participants will be in the study for approx. 21 days. Each participant will have 5 visits to the clinic, with an overnight stay at both dosing visits. Participants will have a number of tests, and they will have to give blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 64 years (both inclusive) at the time of signing informed consent.
* Type 1 diabetes mellitus (as diagnosed clinically) for 12 months or longer.
* Body mass index 18.5 - 28.0 kg/sqm (both inclusive).
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for 12 months or longer.

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening.
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily).
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to 30 min | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum

SECONDARY OUTCOMES:
Continuous subcutaneous infusion related time from bolus to 50% of max insulin aspart concentration | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related time from bolus to max insulin aspart concentration | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to 15 min. | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to 1 hour | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to 1,5 hour | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to 2 hours | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 0 to first time the curve is back to baseline | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related area under the insulin aspart curve, baseline corrected and based on concentrations from 2 hours to first time the curve is back to baseline | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related time from bolus to late 50% of max insulin aspart concentration | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on plasma insulin measured in serum
Continuous subcutaneous infusion related time from bolus to max baseline corrected insulin aspart concentration | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related time from bolus administration to 50% of max baseline corrected Glucose Infusion Rate | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration measured at 56 times during 24 hours
  Calculated based on insulin aspart measured in serum
Continuous subcutaneous infusion related time from bolus administration to max of baseline corrected Glucose Infusion Rate | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 0 to 30 min | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 0 to 1 hour | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 0 to 1,5 hour | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 0 to 2 hours | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 0 to first time the curve is back to baseline | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related area under the glucose infusion rate curve, baseline corrected and based on concentrations from 2 hours to first time the curve is back to baseline | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Area under the glucose infusion rate curve based on concentrations from -2 to 0 hours | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Area under the glucose infusion rate curve based on concentrations from 12 to 14 hours | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related max of baseline corrected Glucose Infusion Rate | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Continuous subcutaneous infusion related time from bolus to late 50% of max baseline corrected glucose infusion rate | Day of dosing: day 1 visit 2, day 1 visit 3 (7-14 days after day 2 of visit 2), based on concentration recorded approximately 57 times during 24 hours
  Calculated based on glucose infusion
Number of adverse events ( AEs) | Day 1-21
  Count of events
Number of hypoglycaemic episodes | Day 1-21
  Count of episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com